CLINICAL TRIAL: NCT03277274
Title: A Phase 1, Non-Randomized, Open-Label Trial to Evaluate the Effect of Hepatic Impairment on the Single Dose Pharmacokinetics of Intravenous TAK-954
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on the Single Dose Pharmacokinetics (PK) of Intravenous TAK-954
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-954-1006; 2017-000714-37 (EudraCT Number); U1111-1196-9190 (Registry Identifier: WHO)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 Mild Hepatic Impairment: TAK-954 0.2 mg (Experimental): TAK-954 0.2 milligram (mg), intravenous, administered as 60-minute infusion, once on Day 1.
  Interventions: Drug: TAK-954
- Group 2 Moderate Hepatic Impairment: TAK-954 0.2 mg (Experimental): TAK-954 0.2 mg, intravenous, administered as 60-minute infusion, once on Day 1.
  Interventions: Drug: TAK-954
- Group 3 Severe Hepatic Impairment: TAK-954 0.2 mg (Experimental): TAK-954 0.2 mg, intravenous, administered as 60-minute infusion, once on Day 1.
  Interventions: Drug: TAK-954
- Group 4 Healthy Participants: TAK-954 0.2 mg (Experimental): TAK-954 0.2 mg, intravenous, administered as 60-minute infusion, once on Day 1.
  Interventions: Drug: TAK-954

INTERVENTIONS:
Drug: TAK-954 — TAK-954 intravenous infusion.

SUMMARY:
The purpose of this study is to evaluate the effect of varying degrees of hepatic function on the single dose PK of IV TAK-954.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. This study will evaluate the safety and tolerability of single intravenous doses of TAK-954 in participants with varying degrees of hepatic function.

The study will enroll approximately up to 32 participants. Participants will be enrolled in one of the 4 treatment groups based on their degree of hepatic impairment which will be determined based on Child-Pugh Score as follow:

* Group 1 TAK-954 0.2 mg: Mild Hepatic Impairment (Child Pugh Class A)
* Group 2 TAK-954 0.2 mg: Moderate Hepatic Impairment (Child Pugh Class B)
* Group 3 TAK-954 0.2 mg: Severe Hepatic Impairment (Child Pugh Class C)
* Group 4 TAK-954 0.2 mg: Healthy Participants

The Child-Pugh classification will assess the severity of 5 hepatic parameters (total serum bilirubin, serum albumin, prothrombin time, ascites and encephalopathy grade) on a scale of 1 (none) to 3 (moderate). Total hepatic impairment score ranges from 5 (mild) to 15 (severe) where higher score indicates more severity.

All participants will receive a single dose of TAK-954 0.2 mg on Day 1.

This study may have a full study design, where Group 1 to Group 4 will enroll approximately 8 participants in each group or a reduced study design, where no participants will be enrolled in Group 1 and approximately 8 participants will be enrolled in Group 2 to Group 4.

This multi-center trial will be conducted in Czech Republic and Slovakia. The overall time to participate in this study is approximately 7 weeks. Participants will remain confined to the clinic for 4 days, with 2 further out-patient visits, and will make a final visit to the clinic 10-14 days after receiving their last dose of TAK-954 for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants (non-childbearing potential), with a body mass index (BMI) between 18 to 35 kilogram per square meter (kg/m^2) (All participants).
2. Participants with hepatic impairment who are medically stable as determined by the investigator, based on medical history and clinical evaluations including physical examinations, clinical laboratory tests, vital sign measurements, and 12-lead ECGs performed at the Screening Visit and at check-in on Day -1 (Group 1 to 3).
3. Healthy participants (Group 4).

Exclusion Criteria:

Participants who have:

1. A history of hepatic carcinoma, hepatorenal syndrome, or presence of a liver mass by ultrasound, CT or MRI, or acute liver disease caused by an infection or drug toxicity (Group 1 to 3).
2. Have severe hepatic encephalopathy ([greater than] > Grade II Portal Systemic Encephalopathy Score) (Group 1 to 3).
3. Surgical porto-systemic shunts, including transjugular intrahepatic portosystemic shunt (Group 1 to 3).
4. A history of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than 1 month prior to trial entry (Group 1 to 3).
5. Bilirubin levels above 5 times the upper limit of normal (ULN) at screening or Day -1 for Groups 1 and 2, there is no limit for Group 3.
6. Severe/advanced ascites and/or pleural effusion which requires emptying and albumin supplementation, as judged by the investigator (Group 1 to 3).
7. Renal creatinine clearance (CLcr) less than or equal to (<=) 50 milliliter per minute (mL/min), calculated using the Cockcroft-Gault equation from the serum creatinine measurement taken at screening (Group 1 to 3).
8. Who have a history of clinically significant endocrine, gastrointestinal (GI) (including motility disorder and intestinal obstruction), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases will be excluded from the trial (Group 4).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- PRA CZ, s.r.o, Prague, Prague, Czechia
- Summit Center of Clinical Research, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Czech Republic and Slovakia from 09 November 2017 to 10 September 2018.
Pre-assignment Details: Participants with normal hepatic function and hepatic impairment were enrolled in 1 of the groups:B(moderate), C(severe) or D(healthy) to receive TAK-954 0.2mg. Based on available safety and PK data from Group B, participants were enrolled in reduced study design and were not enrolled in GroupA(mild). Groups A-D are equal to Groups 1-4 in protocol.
Groups:
- Healthy Participants: TAK-954 0.2 mg: TAK-954 0.2 milligram (mg), infusion, intravenously, once on Day 1.
- Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg; Group C, Severe Hepatic Impairment: TAK-954 0.2 mg: TAK-954 0.2 mg, infusion, intravenously, once on Day 1.
Period: Overall Study
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Started | 8 | 10 | 7
Completed | 8 | 10 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all participants who were enrolled and received the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg | Total
Number analyzed (Participants) | 8 | 10 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.46) | 55.6 (12.25) | 57.9 (12.88) | 57.2 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 5 | 6 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 10 | 7 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 10 | 7 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czech Republic | 3 | 3 | 2 | 8
  Slovakia | 5 | 7 | 5 | 17
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 89.95 (17.098) | 86.77 (19.823) | 87.19 (21.331) | 87.90 (18.667)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 31.1 (3.18) | 30.4 (5.02) | 27.9 (6.18) | 29.9 (4.87)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 169.8 (11.30) | 168.0 (10.47) | 176.1 (6.28) | 170.8 (10.01)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-954 (Total and Free)
Time Frame: Day 1 pre-infusion and at multiple time points (up to 96 hours) post-infusion
Population: The pharmacokinetic (PK) set consisted of all participants who were enrolled and received the correct dose of study drug and had at least 1 measurable plasma concentration or amount of drug in the urine for TAK-954.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 8 | 7
nanogram per milliliter (ng/mL)
  TAK-954 (Total) | 2.629 (19.1) | 2.440 (25.3) | 1.893 (35.4)
  TAK-954 (Free) | 0.1381 (15.6) | 0.1799 (24.4) | 0.1778 (23.1)
Statistical Analysis 1: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — TAK-954 (Total): An analysis of variance (ANOVA) were performed on log transformed Cmax (total TAK-954) to compare each hepatically impaired group with the normal hepatic function group; p = 0.579, ANOVA
Statistical Analysis 2: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group C, Severe Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — TAK-954 (Total): An ANOVA were performed on log transformed Cmax (total TAK-954) to compare each hepatically impaired group with the normal hepatic function group; p = 0.026, ANOVA
Statistical Analysis 3: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — TAK-954 (Free): An ANOVA were performed on log transformed Cmax (Free TAK-954) to compare each hepatically impaired group with the normal hepatic function group; p = 0.020, ANOVA
Statistical Analysis 4: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group C, Severe Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — [test comment as in outcome 1, analysis 3]; p = 0.031, ANOVA

2. Primary Outcome: AUClast: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-954 (Total and Free)
Time Frame: Day 1 pre-infusion and at multiple time points (up to 96 hours) post-infusion
Population: The PK set consisted of all participants who were enrolled and received the correct dose of study drug and had at least 1 measurable plasma concentration or amount of drug in the urine for TAK-954.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 8 | 7
hour*nanogram per milliliter (h*ng/mL)
  TAK-954 (Total) | 28.57 (19.2) | 23.57 (26.2) | 20.19 (32.7)
  TAK-954 (Free) | 1.501 (12.0) | 1.737 (23.0) | 1.898 (19.3)
Statistical Analysis 1: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — TAK-954 (Total): An ANOVA were performed on log transformed AUClast (Total TAK-954) to compare each hepatically impaired group with the normal hepatic function group; p = 0.151, ANOVA
Statistical Analysis 2: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group C, Severe Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.017, ANOVA
Statistical Analysis 3: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — TAK-954 (Free): An ANOVA were performed on log transformed AUClast (Free TAK-954) to compare each hepatically impaired group with the normal hepatic function group; p = 0.129, ANOVA
Statistical Analysis 4: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group C, Severe Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — [test comment as in outcome 2, analysis 3]; p = 0.023, ANOVA

3. Primary Outcome: AUC∞: Area Under the Concentration-time Curve From Time 0 to Infinity for TAK-954 (Total and Free)
Time Frame: Day 1 pre-infusion and at multiple time points (up to 96 hours) post-infusion
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 8 | 7
h*ng/mL
  TAK-954 (Total) | 31.30 (20.1) | 25.44 (27.1) | 22.60 (34.3)
  TAK-954 (Free) | 1.643 (13.8) | 1.875 (24.0) | 2.122 (21.8)
Statistical Analysis 1: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — TAK-954 (Total): An ANOVA were performed on log transformed AUCinf (Total TAK-954) to compare each hepatically impaired group with the normal hepatic function group; p = 0.138, ANOVA
Statistical Analysis 2: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group C, Severe Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.029, ANOVA
Statistical Analysis 3: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — TAK-954 (Free): An ANOVA were performed on log transformed AUCinf (Free TAK-954) to compare each hepatically impaired group with the normal hepatic function group; p = 0.201, ANOVA
Statistical Analysis 4: Comparison: Healthy Participants: TAK-954 0.2 mg vs Group C, Severe Hepatic Impairment: TAK-954 0.2 mg; Test type: Other — [test comment as in outcome 3, analysis 3]; p = 0.023, ANOVA

4. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Time Frame: Up to 14 days after the last dose of study drug (Day 15)
Population: The safety set consisted of all participants who were enrolled and received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 10 | 7
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Markedly Abnormal Electrocardiograms (ECGs)
Time Frame: Up to 14 days after the last dose of study drug (Day 15)
Population: The safety set consisted of all participants who were enrolled and received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 10 | 7
Participants | 0 | 0 | 2

6. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Vital Signs
Time Frame: Up to 14 days after the last dose of study drug (Day 15)
Population: The safety set consisted of all participants who were enrolled and received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 10 | 7
Participants | 0 | 1 | 1

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Values
Time Frame: Up to 14 days after the last dose of study drug (Day 15)
Population: The safety set consisted of all participants who were enrolled and received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 10 | 7
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 30 days after last dose of study drug (Day 31)
Population: The safety set consisted of all participants who were enrolled and received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
Number analyzed (Participants) | 8 | 10 | 7
Participants | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug and no more than 30 days (Day 31) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Healthy Participants: TAK-954 0.2 mg | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 2/8 | 3/10 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants: TAK-954 0.2 mg (N=8) | Group B, Moderate Hepatic Impairment: TAK-954 0.2 mg (N=10) | Group C, Severe Hepatic Impairment: TAK-954 0.2 mg (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT03277274/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03277274/SAP_001.pdf